CLINICAL TRIAL: NCT04816864
Title: Safety and Efficacy of HIs Bundle Pacing Validated by electrophySiological STudy, autonOmic Tests and extRacardiac Vagal Nerve Stimulation (HIS-STORY)
Brief Title: Safety and Efficacy of His Bundle Pacing Validated by Extracardiac Vagal Nerve Stimulation
Acronym: HIS-STORY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: 4th Military Clinical Hospital with Polyclinic, Poland (Other)
Collaborators: Subcarpathian Center for Cardiovascular Intervention (Unknown); Mazovian Speciality Hospital (Unknown); Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Krystian Josiak, Krystian Josiak, MD, PhD, 4th Military Clinical Hospital with Polyclinic, Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4thMilitaryH
Record Dates: First submitted 2021-03-21; First posted 2021-03-25 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Permanent His Bundle Pacing; Permanent Left Bundle Branch Pacing
Keywords: His bundle pacing; left bundle branch pacing; extracardiac vagal nerve stimulation
MeSH Terms: interventions — Electrophysiologic Techniques, Cardiac

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECANS started from the right vagus nerve (Active Comparator): superior ECANS and ultrasonography guided inferior ECANS
  Interventions: Diagnostic Test: extracardiac vagal nerve stimulation (ECANS) + EPS
- ECANS started from the left vagus nerve (Active Comparator): superior ECANS and ultrasonography guided inferior ECANS
  Interventions: Diagnostic Test: extracardiac vagal nerve stimulation (ECANS) + EPS

INTERVENTIONS:
Diagnostic Test: extracardiac vagal nerve stimulation (ECANS) + EPS — The study intervention will consist of 3 steps, all of which will be performed under general anesthesia:
  1. EPS with the measurement of parameters of atrioventricular conduction and programmed atrial and ventricular pacing.
  2. ECANS of the right and the left vagus nerve (from the right and left internal jugular vein, respectively; patients will be randomized to start from the right or the left side) performed during: 1) the patient's spontaneous heart rhythm (if present); 2) HB/LBB pacing with permanently programmed impulse parameters; 3) HB/LBB pacing at a pacing threshold of +0.1 V; and 4) 5 minutes after intravenous injection of atropine (0.02-0.04 mg/kg).
  3. EPS with the measurement of parameters of atrioventricular conduction and programmed atrial and ventricular pacing.

SUMMARY:
Different studies for extracardiac vagal nerve stimulation (ECANS) have been published and confirmed the influence of the vagus nerve on automaticity and conduction properties of the sinus node, atria, atrioventricular node, as well as the His-Purkinje system (HPS) and ventricles. However, there are limited data on the clinical value and impact of ECANS as well as vagus nerve activity on the parameters of permanent His-bundle (HB) or left bundle branch (LBB) pacing. Moreover, there have been no prospective studies evaluating the feasibility and efficacy of ECANS and the management of ECANS-induced scenarios, such as an exit block, increase in pacing threshold, as well as vagally mediated arrhythmias and conduction abnormalities in patients with physiological conduction system pacing (HB/LBB pacing).

The objective of the HIS-STORY study in humans is to evaluate the clinical value of ECANS in patients with HB/LBB pacing for further development of patient-centered management strategy.

DETAILED DESCRIPTION:
This is a multicenter, prospective, open-label, randomized, interventional study enrolling patients with indications for permanent cardiac pacing according to the current European Society of Cardiology Guidelines on Cardiac Pacing. All participants will undergo permanent pacemaker implantation for HB or LBB pacing. Subsequently, an invasive electrophysiological study (EPS) and ECANS will be performed. The 2 x 2 randomisation will be performed, i.e. right vs left side superior ECANS and blinded for operator ultrasonography guided effective vs ineffective inferior vagal nerve stimulation). The randomisation will prove the feasibility and efficacy of superior ECANS and feasibility, efficacy, and reproducibility of ultrasonography guided inferior ECANS. All the measured parameters as well as demographic and clinical data will be recorded in the study database. Patients with an exit block or an increase in a pacing threshold of an HB/LBB electrode will be further managed by electrophysiologists from the research group. The management will be based on clinical assessment and patient's decision and may involve pacemaker reprogramming, pacemaker upgrade with a back-up pacing electrode implantation, or cardio-neuro-ablation.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent form
* effective and stable HB or LBB pacing
* sinus rhythm during the intervention procedure

Exclusion Criteria:

* contraindications to invasive EPS
* contraindications to general anesthesia
* contraindications to atropine administration (e.g., glaucoma)
* persistent atrial fibrillation or atrial flutter
* pregnancy
* diseases that may cause autonomic system neuropathy
* use of medications that may affect the parasympathetic system
* a history of cardiac surgery
* a history of ablation due to arrhythmia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-02 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Loss of HB/LBB capture or significant increase in pacing threshold | 0-12 months after HB/LBB pacemaker implantation
  significant increase in pacing threshold = above the permanently programmed impulse amplitude of HB/LBB electrode induced by ECANS

SECONDARY OUTCOMES:
A nonsignificant increase in pacing threshold | 0-12 months after HB/LBB pacemaker implantation
  below the permanently programmed impulse amplitude of HB/LBB electrode induced by ECANS
Prolongation of the stimulus-QRS interval during HB/LBB pacing induced by ECANS | 0-12 months after HB/LBB pacemaker implantation

OTHER OUTCOMES:
Any arrhythmia induced by ECANS | 0-12 months after HB/LBB pacemaker implantation

CONTACTS AND LOCATIONS:
Overall Officials: Krystian Josiak, MD, PhD, Principal Investigator — 4th Military Clinical Hospital with Polyclinic, Poland
Locations (3):
- Poland (3):
  - 4th Military Hospital, Cardiology Department, Wroclaw, Lower Silesian Voivodeship
  - Mazovian Speciality Hospital, Cardiology Department, Radom, Masovian Voivodeship
  - Subcarpathian Center for Cardiovascular Intervention, Sanok, Podkarpackie Voivodeship

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abdelrahman M, Subzposh FA, Beer D, Durr B, Naperkowski A, Sun H, Oren JW, Dandamudi G, Vijayaraman P. Clinical Outcomes of His Bundle Pacing Compared to Right Ventricular Pacing. J Am Coll Cardiol. 2018 May 22;71(20):2319-2330. doi: 10.1016/j.jacc.2018.02.048. Epub 2018 Mar 10. PMID 29535066
- [Result] Kronborg MB, Mortensen PT, Poulsen SH, Gerdes JC, Jensen HK, Nielsen JC. His or para-His pacing preserves left ventricular function in atrioventricular block: a double-blind, randomized, crossover study. Europace. 2014 Aug;16(8):1189-96. doi: 10.1093/europace/euu011. Epub 2014 Feb 7. PMID 24509688
- [Result] Dandamudi G, Vijayaraman P. How to perform permanent His bundle pacing in routine clinical practice. Heart Rhythm. 2016 Jun;13(6):1362-6. doi: 10.1016/j.hrthm.2016.03.040. Epub 2016 Mar 22. No abstract available. PMID 27016475
- [Result] Josiak K, Nowak K, Fuglewicz A, Jagielski D, Banasiak W, Ponikowski P. Does right ventricular pacing increase the risk of ventricular arrhythmias in patients with an implantable cardioverter-defibrillator? Kardiol Pol. 2014;72(4):381-4. doi: 10.5603/KP.2014.0073. No abstract available. PMID 24733700
- [Result] Sharma PS, Dandamudi G, Naperkowski A, Oren JW, Storm RH, Ellenbogen KA, Vijayaraman P. Permanent His-bundle pacing is feasible, safe, and superior to right ventricular pacing in routine clinical practice. Heart Rhythm. 2015 Feb;12(2):305-12. doi: 10.1016/j.hrthm.2014.10.021. Epub 2014 Oct 22. PMID 25446158
- [Result] Burri H, Jastrzebski M, Vijayaraman P. Electrocardiographic Analysis for His Bundle Pacing at Implantation and Follow-Up. JACC Clin Electrophysiol. 2020 Jul;6(7):883-900. doi: 10.1016/j.jacep.2020.03.005. PMID 32703577
- [Result] Zysko D, Gajek J, Kozluk E, Mazurek W. Electrocardiographic characteristics of atrioventricular block induced by tilt testing. Europace. 2009 Feb;11(2):225-30. doi: 10.1093/europace/eun299. Epub 2008 Nov 5. PMID 18987129
- [Result] Klank-Szafran M, Stec S, Sledz J, Janion M. [Radiofrequency ablation and cardioneuroablation for AVNRT and atrioventricular block]. Kardiol Pol. 2010 Jun;68(6):720-4. Polish. PMID 20806214
- [Result] Pachon JC, Pachon EI, Pachon JC, Lobo TJ, Pachon MZ, Vargas RN, Jatene AD. "Cardioneuroablation"--new treatment for neurocardiogenic syncope, functional AV block and sinus dysfunction using catheter RF-ablation. Europace. 2005 Jan;7(1):1-13. doi: 10.1016/j.eupc.2004.10.003. PMID 15670960
- [Result] Stec S, Dobaj L, Sledz A, Stepien-Walek AM, Ton V, Sledz J. Cardioneuroablation for management of cardioinhibitory vasovagal syncope and pacemaker complications. HeartRhythm Case Rep. 2020 May 11;6(8):531-534. doi: 10.1016/j.hrcr.2020.04.021. eCollection 2020 Aug. No abstract available. PMID 32817835